CLINICAL TRIAL: NCT00915564
Title: A Phase I, Open-Label, Single-Sequence Drug-Drug Interaction Trial in Subjects On Stable Methadone Maintenance Therapy, to Investigate the Potential Pharmacokinetic Interaction Between TMC435 and Methadone, at Steady-State
Brief Title: A Study to Investigate the Potential Pharmacokinetic Interaction Between TMC435 and Methadone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015934; TMC435-TIDP16-C110 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; HCV; Hepatitis C Virus; HCV negative; Protease inhibitor; Methadone; TMC435
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC435 + methadone (Experimental): Supervised intake of individualized methadone dose (range, 30 to 150 mg once daily) from Day -14 to Day -1; followed by addition of 150 mg dose of TMC435 once daily from Day 1 to Day 7 along with methadone; and later followed by continued intake of individualized methadone 30 to 32 days follow-up.
  Interventions: Drug: TMC435; Other: Methadone

INTERVENTIONS:
Drug: TMC435 — Participants will receive 150 mg dose of TMC435 orally (by mouth) once daily for 7 days of treatment (from Day 1 to Day 7).
Other: Methadone — Participants will receive supervised individualized methadone dose (dose of methadone will be adjusted for each participant between a range of 30 and 150 mg daily [extremes included]) from Day -14 untill Day 8. Participants will continue to receive individualized methadone during follow up of 30 to 32 days.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state (constant concentration of medication in the blood) TMC435 (150 mg, once a day) on the steady state pharmacokinetics (what the body does to the medication) of R- and S-methadone.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention) drug-drug interaction (TMC435 versus methadone) study. Approximately 12 hepatitis C virus-negative opioid-dependent participants on stable maintenance therapy (for at least 30 days before screening) will be enrolled in the study. The study will consist of 3 phases: 1) Run-in phase: during this phase, participants will take individualized (dose of methadone will be adjusted for each participant between a range of 30 and 150 mg daily) dose of methadone from Day -14 (14 days before the first intake of TMC435) till Day -1 (1 day before the first intake of TMC435), which will be supervised by the medical staff. 2) 7 days treatment phase: during this phase, the participants will take 150 mg dose of TMC435 once daily from Day 1 to Day 7 orally (by mouth) plus the individualized dose of methadone which will be supervised by the medical staff. 3) Follow-up phase: during this phase, the participants will continue to take only the individualized dose of methadone for 30-32 days. Safety evaluations will include assessment of adverse events, clinical laboratory tests, cardiovascular safety, physical examination and alcohol breath test. The total study duration will be of 22 days excluding screening and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Receiving once daily oral methadone maintenance therapy at a stable individualized dose of 30 to 130 mg once daily for at least 30 days prior to screening
* Agreeing not to change the current methadone dose from screening until Day7 included and to have a daily observed and documented methadone intake from Day-14 until Day8 and to have a daily observed and documented TMC435 intake from Day1 until Day 7
* Having obtained approval from his/her addiction physician for participation in the trial and addiction physician agrees to provide medical care for the volunteer after discharge from the testing facility

Exclusion Criteria:

* No female of childbearing potential, except if using effective birth control methods during the trial and for at least 30 days after the end of the treatment period
* No positive testing for drugs of abuse
* No positive testing for Hepatitis A, B and C and for HIV1 and 2
* Impaired liver disease or other clinically relevant diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Predose plasma concentration of S-methadone | Day -4 to Day 6
Maximum plasma concentration of S-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Minimum plasma concentration between 0 hour and dosing interval of S-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Average steady-state plasma concentration of S-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Time to reach the maximum plasma concentration of S-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Area under the curve from time of administration up to 24 hours post dosing of S-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Fluctuation index of S-methadone, ie, percentage fluctuation (variation between maximum and minimum concentration at steady-state) | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Predose plasma concentration of R-methadone | Day -4 to Day 7
Maximum plasma concentration of R-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Minimum plasma concentration between 0 hour and dosing interval of R- and S-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Average steady-state plasma concentration of R-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Time to reach the maximum plasma concentration of R-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Area under the curve from time of administration up to 24 hours post dosing of R-methadone | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Fluctuation index of R-methadone, ie, percentage fluctuation (variation between maximum and minimum concentration at steady-state) | On Day -1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose
Predose plasma concentration of TMC435 | Day 4 to Day 6
Maximum plasma concentration of TMC435 | On Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose and on Day 8 at 24 hour postdose
Minimum plasma concentration between 0 hour and dosing interval of TMC435 | On Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose and on Day 8 at 24 hour postdose
Average steady-state plasma concentration of TMC435 | On Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose and on Day 8 at 24 hour postdose
Time to reach the maximum plasma concentration of TMC435 | On Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose and on Day 8 at 24 hour postdose
Area under the curve from time of administration up to 24 hours post dosing of TMC435 | On Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose and on Day 8 at 24 hour postdose
Fluctuation index of TMC435, ie, percentage fluctuation (variation between maximum and minimum concentration at steady-state) | On Day 7 at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours postdose and on Day 8 at 24 hour postdose

SECONDARY OUTCOMES:
Short Opiate Withdrawal Scale Scores | On Day-1 and Day 7 at 2 hour and 4 hour predose; on Day-7, Day-2, and Day 1 to Day 6 at predose
  Short Opiate Withdrawal Scale is used for the assessment of opioid withdrawal. It consists of 10 items and items are designed to measure symptoms, on a scale from 0 to 3 (0= None, 1= Mild, 2= Moderate, 3= Severe). The total score ranges from 0 (best) to 30 (worst). Higher scores indicate worsening.
Desires for Drugs Questionnaire | On Day-1 and Day 7 at 2 hour and 4 hour predose; on Day-7, Day-2, and Day 1 to Day 6 at predose
Resting pupil diameter | On Day-1 and Day 7 at 2 hour and 4 hour predose; on Day-7, Day-2, and Day 1 to Day 6 at predose
  Pupillometry will be performed and resting pupil diameter will be assessed with a validated pupillograph.
Number of participants with adverse events as a measure of safety and tolerability | Up to 30 to 32 days after the last medication dose

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (1):
- Toronto, Canada

REFERENCES:
- See also: A Phase I, Open-Label, Single-Sequence Drug-Drug Interaction Trial in Subjects On Stable Methadone Maintenance Therapy, to Investigate the Potential Pharmacokinetic Interaction Between TMC435 and Methadone, at Steady-State — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1020&filename=CR015934_CSR.pdf